CLINICAL TRIAL: NCT05924542
Title: The Smart Way to Beat Stress at Work - SOMA
Brief Title: Kelaa Mental Resilience App for Employees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wuerzburg (Other)
Collaborators: SOMA Analytics UK (Unknown)
Responsible Party: Principal Investigator, Dr. Silvana Weber, Lead Researcher, University of Wuerzburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H2020-725832
Record Dates: First submitted 2023-05-25; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Stress; Presenteeism; Absenteeism

STUDY DESIGN:
Intervention Model Description: RCT with intervention and wait-list control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants had access to the Kelaa Mental Resilience App for 4 weeks. Thus, participants in the intervention group could complete a maximum of 28 sessions and track a maximum of 28 nights. It was completely left to the user to what extent s/he wanted to engage with the app. The app seeks to translate insights from scientific research on psychology, sleep medicine, and neuroscience into an action-based program. It draws on the tenets of clinical, health, positive, cognitive, biological, and social psychology to foster recovery and growth. "Kelaa" aims to reduce stress and increase well-being of the user, specifically in the workplace. Users learn new behaviors and best practices through different means, for example, based on CBT and mindfulness based cognitive therapy. The app is designed to implement lifestyle changes through (1) measuring behavior, cognitions, and emotions (tracking module) and (2) providing psycho-educational content (intervention module).
  Interventions: Behavioral: Kelaa Mental Resilience App
- Wait-list Control Group (No Intervention): Participants in the waitlist control group received no intervention and no tracking opportunity for the duration of the trial (6 weeks), yet they had unrestricted access to treatment as usual within their companies. Upon completion of the trial, participants in the waitlist control group received access to the "Kelaa" app.

INTERVENTIONS:
Behavioral: Kelaa Mental Resilience App — Users can track their stress, wellbeing, and resilience via short in-app questionnaires. The app uses inbuilt sensors in smartphones to measure sleep quality and quantity. Personalized feedback on questionnaire scores and on sleep data are given. Users access structured science-based content on factors contributing to reduced stress and improved well-being. "Kelaa" provides the user with evidence-based interventions grounded in current research, e.g., from sleep science and psychology. Users can choose from a variety of topics, based on their results from the tracking module and personal interest, and then journey through the self-selected goals. Each goal includes six to seven "daily sessions", aiming to increase personal resources by providing information, exercises, and reflection. During each daily session, relevant research and expected benefits are outlined, before users are instructed, e.g., in specific stress management and resilience techniques, to encourage behavior change.
  Arms: Intervention Group

SUMMARY:
The goal of this randomized control trial is to detect and prevent work-related psychological stress among European workers early on, aiming to mitigate its adverse health consequences, including burnout and depression. Soma Analytics has developed a smartphone-based system that comprises a diagnostic module utilizing smartphone sensors to collect and analyze stress biomarkers and an interventional module to reduce stress levels. The main questions this study aims to answer are:

* Hypothesis 1: Compared to the waitlist control, after using the app for 4 weeks, participants in the app group will report (a) lower levels of stress (cognitive and general), (b) higher levels of wellbeing, (c) higher levels of resilience, and (d) fewer sleeping troubles.
* Hypothesis 2: The observed effects will be more intense the more the user interacts with the app throughout the duration of the study.

Participants (employees from six organizations in three European countries) will use the app for 4 weeks. Their levels of stress, well-being, resilience, and sleeping troubles are assessed at baseline, after 2 weeks (mid-intervention), 4 weeks (end of intervention), and 6 weeks (follow-up).

Researchers will compare the intervention group with the waitlist control group to see if levels of stress, well-being, resilience, and sleeping troubles change over time.

DETAILED DESCRIPTION:
Work-related psycho-social risks and stress have a significant impact on numerous workplaces in Europe, leading to adverse health and business outcomes, as previous research has shown. Prolonged stress have been shown to eventually result in burnout and depression. In 2013, the total annual cost of work-related stress and depression in the EU-27 was estimated to be €617 billion. This figure encompasses expenses borne by employers due to absenteeism (€272 billion), reduced productivity (€242 billion), healthcare costs (€63 billion), and social welfare expenses (€39 billion).

The primary objective of the project is to identify and prevent work-related psychological stress that can lead to negative health outcomes like burnout and depression. To achieve this, Soma Analytics has developed a comprehensive smartphone-based system that promotes mental resilience by continuously monitoring well-known stress biomarkers. The solution consists of three modules: a diagnostic module that utilizes smartphone sensors to gather and analyse stress biomarkers, an interventional module comprising smartphone apps aimed at reducing stress levels, and an analytics module that aggregates anonymous data to identify specific human resources issues, such as abnormal stress levels in particular departments. Soma's approach to preventing stress and promoting positive mental health in the workplace includes validated psychological interventions that are tailored to each individual, guiding users through a personalized micro-learning journey. The extensive database of interventions covers a wide range of topics, providing diverse options for users.

This large-scale randomized controlled trial (RCT) involves participants from six organizations across three European countries. It is conducted to validate the solution's effectiveness in reducing stress and improving overall well-being. In a real-world work environment, the investigators examine the effectiveness of Soma's solution. It was hypothesized that it may reduce stress levels, enhance overall well-being, boost resilience, and reduce sleep difficulties compared to a waitlist control group.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old
* Having a mobile phone with internet access
* Accepting informed consent
* Being employed in one of the participating organizations at the time of the recruitment

Exclusion Criteria:

* Younger than 18
* Being unemployed at the time of recruitment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 678 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

PRIMARY OUTCOMES:
Change in General and Cognitive Stress | at baseline (T1, week 0), mid-intervention (T2, week 2), end-intervention (T3, week 4), and two-week follow-up (T4, week 6).
  Self-reported levels of stress were assessed with the two subscales General Stress (four items, e.g., "How often have you been stressed?") and Cognitive Stress (four items, e.g., "How often have you had problems concentrating?") from the Copenhagen Psychosocial Questionnaire - Revised Version (COPSOQ II; Pejtersen et al., 2010).The items were answered on a five-point scale (1 = not at all; 2 = a small part of the time; 3 = part of the time; 4 = a large part of the time; 5 = all the time). Higher values indicate more stress.

SECONDARY OUTCOMES:
Change in Wellbeing | at baseline (T1, week 0), mid-intervention (T2, week 2), end-intervention (T3, week 4), and two-week follow-up (T4, week 6).
  Subjective wellbeing was measured with the Warwick-Edinburgh Mental Wellbeing Scale (Tennant et al., 2007). Seven items (e.g., "I've been feeling relaxed.") were answered on a five-point scale (1 = none of the time; 2 = rarely; 3 = some of the time; 4 = often; 5 = all of the time). Higher values indicate more wellbeing.
Change in Resilience | at baseline (T1, week 0), mid-intervention (T2, week 2), end-intervention (T3, week 4), and two-week follow-up (T4, week 6).
  We assessed resilience with the 13-item Resilience Scale (RS-13; Leppert et al., 2008), a short form of the Resilience Scale (RS-25; Wagnild and Young, 1993). Items (e.g., "I usually take things in stride.") were answered on a seven-point scale (1 = strongly disagree to 7 = strongly agree). Higher values indicate more resilience.
Change in Sleeping Troubles | at baseline (T1, week 0), mid-intervention (T2, week 2), end-intervention (T3, week 4), and two-week follow-up (T4, week 6).
  Participants were asked about sleeping troubles with the subscale Sleeping Troubles from the COPSOQ II (Pejtersen et al., 2010). Four items (e.g., "How often have you slept badly and restlessly?") were answered on a five-point scale (1 = not at all; 2 = a small part of the time; 3 = part of the time; 4 = a large part of the time; 5 = all the time). Higher values indicate more sleeping troubles.
Change in Social Community at Work | at baseline (T1, week 0), mid-intervention (T2, week 2), end-intervention (T3, week 4), and two-week follow-up (T4, week 6).
  Participants indicated their sense of cooperation and social community at work with the subscale Social Community at Work from the COPSOQ II (Pejtersen et al., 2010). Three items (e.g., "Do you feel part of a community at your place of work?") were answered on a five-point scale (1 = not at all; 2 = a small part of the time; 3 = part of the time; 4 = a large part of the time; 5 = all the time). Higher values indicate more sense of social community.
Change in Physical Health Impairment | at baseline (T1, week 0), mid-intervention (T2, week 2), end-intervention (T3, week 4), and two-week follow-up (T4, week 6).
  We assessed participants self-reported physical health levels with the SF-36 Version 2 (Jenkinson et al., 1999). Participants were asked to indicate their agreement to four items (e.g., "Because of your physical health, you were limited in the kind of work or other activities.") on a scale from 1 = none of the time to 5 = all of the time. Higher values indicate worse physical health.
Change in Work productivity and activity impairment | at baseline (T1, week 0), mid-intervention (T2, week 2), end-intervention (T3, week 4), and two-week follow-up (T4, week 6).
  The Work Productivity and Activity Impairment Questionnaire: General Health V2.0 (WPAI:GH; Reilly et al., 1993) asked participants about the impact of health problems on their ability to work and perform regular activities over the past week. Three items (i.e., "During the past 7 days, how many hours did you miss from work because of your health problems?" "…, how many hours did you miss from work because of any other reason, such as vacation, holidays, time off to participate in this study?" "…, how many hours did you actually work?") were provided with open text fields. Two items asked for a rating on a bipolar 11-point scale (e.g., "…, how much did your health problems affect your productivity while you were working?"; 0 = Health problems had no effect on my work to 10 = Health problems completely prevented me from working).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Lorenz, Principal Investigator — SOMA Analytics UK
Locations (1):
- Soma Analytics UK, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The raw data may be made available by the PI or lead researcher, without undue reservation, to any qualified researcher.
Time Frame: The raw data may be made available at any point in time until 10 years after this research has been completed (i.e. until September 2028).
Access Criteria: The raw data may be made available by the PI or lead researcher upon request, without undue reservation, to any qualified researcher.

REFERENCES:
- [Result] Weber S, Lorenz C, Hemmings N. Improving Stress and Positive Mental Health at Work via an App-Based Intervention: A Large-Scale Multi-Center Randomized Control Trial. Front Psychol. 2019 Dec 6;10:2745. doi: 10.3389/fpsyg.2019.02745. eCollection 2019. PMID 31866915
- [Derived] de Miquel C, Moneta MV, Weber S, Lorenz C, Olaya B, Haro JM. The Mediating Role of General and Cognitive Stress on the Effect of an App-Based Intervention on Productivity Measures in Workers: Randomized Controlled Trial. J Med Internet Res. 2023 Jul 3;25:e42317. doi: 10.2196/42317. PMID 37399056